CLINICAL TRIAL: NCT02931734
Title: Analysis of the Association of Products for the Treatment of Cervical Dentin Hypersensitivity
Brief Title: Assessment of Different Protocols for Cervical Dentin Hypersensitivity Treatment
Acronym: CDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE:35634614.2.0000.5152
Record Dates: First submitted 2016-10-03; First posted 2016-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Hypersensitivity Dentin; Dentin Sensitivity; Dentin Hypersensitivity; Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Clinpro Sealant; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Resin modified glass ionomer (RMGI) (Active Comparator): Resin modified glass ionomer; an application every 48 hours; 4 sessions.
  Interventions: Drug: Resin modified glass ionomer
- Potassium Nitrate 2% (KF) (Active Comparator): Potassium Nitrate and Sodium fluoride 2%; an application every 48 hours; 4 sessions.
  Interventions: Drug: Potassium Nitrate 2%
- Low level laser therapy - GaAlAs (LLLT) (Active Comparator): Low level laser therapy - GaAlAs; an application every 48 hours; 4 sessions.
  Interventions: Procedure: Low level laser therapy
- RMGI and KF (Active Comparator): Resin modified glass ionomer and potassium nitrate and sodium fluoride 2%; an application of the two associated products, every 48 hours; 4 sessions.
  Interventions: Drug: Resin modified glass ionomer; Drug: Potassium Nitrate 2%
- RMGI and LLLT (Active Comparator): Resin modified glass ionomer and Low level laser therapy - GaAlAs; an application of the two associated products, every 48 hours; 4 sessions.
  Interventions: Drug: Resin modified glass ionomer; Procedure: Low level laser therapy
- KF and LLLT (Active Comparator): Potassium Nitrate and Sodium fluoride 2% and Low level laser therapy - GaAlAs; an application of the two associated products, every 48 hours; 4 sessions.
  Interventions: Drug: Potassium Nitrate 2%; Procedure: Low level laser therapy
- RMGI, KF, LLLT (Active Comparator): Resin modified glass ionomer, potassium nitrate and sodium fluoride 2% and Low level laser therapy - GaAlAs ; an application of the three associated products, every 48 hours; 4 sessions.
  Interventions: Drug: Resin modified glass ionomer; Drug: Potassium Nitrate 2%; Procedure: Low level laser therapy

INTERVENTIONS:
Drug: Resin modified glass ionomer — Prophylaxis, washing and removing water excess , apply the Clinpro forming a uniform layer of 0.5mm, lightcure for 20 seconds
  Other Names: Clinpro
  Arms: RMGI and KF; RMGI and LLLT; RMGI, KF, LLLT; Resin modified glass ionomer (RMGI)
Drug: Potassium Nitrate 2% — Prophylaxis, apply uniformly on the teeth, wait 10 minutes, remove the gel from the teeth with cotton and abundant water.
  Other Names: Desensibilize KF
  Arms: KF and LLLT; Potassium Nitrate 2% (KF); RMGI and KF; RMGI, KF, LLLT
Procedure: Low level laser therapy — Prophylaxis, applying infrared laser at low power in points: mesial, buccal, distal and in the apical point in the foyer of fornix with power of 110MW for 11 seconds at each point.
  Other Names: Photon Lase III
  Arms: KF and LLLT; Low level laser therapy - GaAlAs (LLLT); RMGI and LLLT; RMGI, KF, LLLT

SUMMARY:
The aim of this study is through a randomized clinical trial, double blind, splith-mouth, evaluate the various types of protocols and clinical efficacy in the reduction or even elimination of dentinal hypersensitivity by the agents Desensibilize KF - FGM Dental Products, Clinpro - 3M Company, Minnesota - USA, Photon Laser III - DMC, Brazil, Desensibilize KF and laser, Desensibilize KF and Clinpro, laser and Clinpro and the association of all products. Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
Cervical dentin hypersensitivity is a painful condition and is a clinical challenge due to different treatment strategies available. The aim of this study is through a randomized clinical trial, double blind, splith-mouth, evaluate the various types of protocols and clinical efficacy in the reduction or even elimination of dentinal hypersensitivity. A hundred forty teeth of healthy patients of both sexes were selected. Visual Analog Scale was used pain (VAS) to measure the intensity of the patient's pain. The teeth will be randomly divided into 7 different groups according to the desensitization treatment under study: Desensibilize KF - FGM Dental Products, Clinpro - 3M Company, Minnesota - USA, Photon Laser III - DMC, Brazil, Desensibilize KF and laser, Desensibilize KF and Clinpro, laser and Clinpro and the association of all products. Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* presence of dentin exposure lesions with clinical diagnosis of moderate or severe tooth sensitivity
* good oral hygiene.

Exclusion Criteria:

* cavities,
* presence of periodontal disease and or parafunctional habits,
* cracks or enamel fractures,
* extensive or unsatisfactory restorations,
* recent restorations involving the labial surface,
* dentures,
* orthodontics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Level of cervical dentin hypersensitivity, measured by visual analog scale | 24 weeks
  Evaluate the reduction in Cervical Dentin Hypersensitivity with a 24 weeks follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo V Soares, PhD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orchardson R, Gangarosa LP Sr, Holland GR, Pashley DH, Trowbridge HO, Ashley FP, Kleinberg I, Zappa U. Dentine hypersensitivity-into the 21st century. Arch Oral Biol. 1994;39 Suppl:113S-119S. doi: 10.1016/0003-9969(94)90197-x. No abstract available. PMID 7702459
- [Background] Lussi A. Erosive tooth wear - a multifactorial condition of growing concern and increasing knowledge. Monogr Oral Sci. 2006;20:1-8. doi: 10.1159/000093343. PMID 16687880
- [Background] Davari A, Ataei E, Assarzadeh H. Dentin hypersensitivity: etiology, diagnosis and treatment; a literature review. J Dent (Shiraz). 2013 Sep;14(3):136-45. PMID 24724135
- [Background] Canadian Advisory Board on Dentin Hypersensitivity. Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. J Can Dent Assoc. 2003 Apr;69(4):221-6. PMID 12662460
- [Background] Coleman TA, Grippo JO, Kinderknecht KE. Cervical dentin hypersensitivity. Part II: Associations with abfractive lesions. Quintessence Int. 2000 Jul-Aug;31(7):466-73. PMID 11203968
- [Background] Brannstrom M. Sensitivity of dentine. Oral Surg Oral Med Oral Pathol. 1966 Apr;21(4):517-26. doi: 10.1016/0030-4220(66)90411-7. No abstract available. PMID 5218158
- [Background] Grippo JO, Simring M, Coleman TA. Abfraction, abrasion, biocorrosion, and the enigma of noncarious cervical lesions: a 20-year perspective. J Esthet Restor Dent. 2012 Feb;24(1):10-23. doi: 10.1111/j.1708-8240.2011.00487.x. Epub 2011 Nov 17. PMID 22296690
- [Background] Grippo JO. Biocorrosion vs. erosion: the 21st century and a time to change. Compend Contin Educ Dent. 2012 Feb;33(2):e33-7. PMID 23268573